CLINICAL TRIAL: NCT00035100
Title: An Open-Label Phase IIa Trial Evaluating the Safety and Efficacy of EPO906 as Therapy in Patients With Advanced Ovarian, Primary Fallopian, or Primary Peritoneal Cancer
Brief Title: EPO906 Therapy in Patients With Advanced Ovarian, Primary Fallopian, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2203
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms
Keywords: ovarian; ovary; peritoneal cancer; fallopian cancer; cancer; tumor; tumour; neoplasm; carcinoma; intravenous; epothilone
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms; Neoplasms; Carcinoma | interventions — epothilone B

ARMS (1):
- EPO906 (Experimental)
  Interventions: Drug: epothilone b

INTERVENTIONS:
Drug: epothilone b
  Other Names: EPO906

SUMMARY:
This study will examine whether the new investigational drug EPO906, given by intravenous infusion (IV directly into the vein), is effective in shrinking tumors and preventing the growth of cells that cause ovarian, fallopian, or peritoneal cancers. Recruitment in the United States is complete but the study is still enrolling in other countries.

ELIGIBILITY:
Inclusion Criteria:

The following patients may be eligible for the study:

* Histologically or cytologically documented evidence of ovarian, primary Fallopian or primary peritoneal cancer with at least one measurable lesion (if previous radiation treatment, the target lesion must have demonstrated progression since the radiation)
* Must have a life expectancy of greater than three (3) months
* Prior failure to respond following front-line treatment with a taxane and platinum (or a combination therapy) may be eligible.

Exclusion Criteria:

The following patients are not eligible for the study:

* Patients with radiation therapy or chemotherapy within the last four weeks
* Patients who have had any chemotherapy not containing a taxane and platinum for their disease
* Patients with borderline ovarian and macropapillary tumors
* Patients with unresolved bowel obstruction
* Patients with symptomatic CNS metastases or leptomeningeal involvement
* Patients with any peripheral neuropathy or unresolved diarrhea greater than Grade 1
* Patients with severe cardiac insufficiency
* Patients taking Coumadin or other warfarin-containing agents with the exception of low dose Coumadin (1 mg or less) for the maintenance of in-dwelling lines or ports
* History of another malignancy within 5 years prior to study entry except curatively treated non-melanoma skin cancer or cervical cancer in situ
* Patients with active or suspected acute or chronic uncontrolled infection including abcesses or fistulae
* HIV+ patients
* Pregnant or lactating females.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2001-09; Primary Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Tumor response rate | Every 2 cycles
  tumor response was defined by the Response Evaluation Criteria in Solid Tumors (RECIST).

SECONDARY OUTCOMES:
Time to disease progression | from start of treatment to documented disease progression, death from study indication, or the date of last follow-up
Overall survival | measured from the start of treatment to the date of death or the last date the patient was known to be alive.
Duration of response | Every 3 months
  duration of response in patients with complete response (CR) or partial response (PR)
recording all adverse events (AEs) and serious adverse events (SAEs) | Every 3 months
  Safety and tolerability of patupilone by monitoring and recording all AEs and SAEs, regular monitoring of hematology, blood chemistry and urine lalues, vital signs, ECG and physical examinations
pharmacogenetic analyses with blood and tumor samples from these patients | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Novartis Investigative Site, New Brunswick, New Jersey, United States
- Novartis Investigative Site, Toronto, Ontario, Canada
- Netherlands (3):
  - Novartis Investigative Site, Enschede, Netherlands
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Zwolle
- Slovakia (2):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
- Novartis Investigative Site, Surrey, United Kingdom